CLINICAL TRIAL: NCT05847907
Title: Comparison of Osstem KS SA Versus KS BA for the Patient With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: RCT KS-SA Versur KS-BA in Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: Melodia, Dario, M.D. (Individual); Pisano, Milena, M.D. (Individual); Dr. Aurea M. I. Lumbau (Unknown); Prof. Silvio Mario Meloni (Unknown); Prof. Edoardo Baldoni (Unknown)
Responsible Party: Principal Investigator, Marco Tallarico, Assistent Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UNISS_PHD_Osstem_6
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Dental Implant; Diabetes
Keywords: Dental Implant; Diabetics Patients; Implant-abutment connection
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: patients, centralized radiographic assessor, outcome assessors, and the statistical advisors will be blind to the used implants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BA Surface test group (Experimental): Common procedures: Implants placement in subjects with type 2 diabetes who have lost at least one tooth element and need of a prosthetic implant-supported rehabilitation.
  Test procedure: use of implant with BA surface in type 2 diabetic patients.
  Interventions: Device: Implant placement
- SA Surface control group (Active Comparator): Common procedures: Implants placement in subjects with type 2 diabetes who have lost at least one tooth element and need of a prosthetic implant-supported rehabilitation. Control procedure: use implant with SA surface in type 2 diabetic patients
  Interventions: Device: Implant placement

INTERVENTIONS:
Device: Implant placement — Implant placement in subject with type 2 diabetes mellitus. Implant placement in subjects with type 2 diabetes mellitus. Implants with BA surface will be placed in one group of subjects and implants with SA surface in the other group.

SUMMARY:
The aim of this randomized controlled trial is to evaluate whether is better to place KS Osstem Implants with BA or SA surface placed in patients with type 2 diabetes, and to compare clinical and radiographic data.

ELIGIBILITY:
Inclusion Criteria:

* - Patients of at least 18 years old able to sign an informed consent.
* Patients with at least a single tooth loss in the maxilla or mandible. Patient will provide only one site for the research. Implant sites must allow the placement of implants of at least 3.5 mm (upper laterals and lower incisors); 4 mm (central incisors, canines, and premolars) or 4.5 (molars) mm of diameter and at least 7 mm of length.
* Smokers will be included and categorized into: 1) non smokers; 2) moderate smokers (smoking up to 10 cigarettes/day); 3) heavy smokers (smoking more than 11 cigarettes/day).
* Patients with a plaque index (PI) of less than, or equal to 25% at the time of surgery.
* In case of post-extractive sites, they must have been healing for at least 4 months before being treated in the study.
* Patients with controlled type 2 diabetes mellitus with a duration of at least 1 years of disease evaluation and baseline glycated hemoglobin A1c (HbA1c) values between 7.5% and 12% at the time of implant placement will be included.

Exclusion Criteria:

* General contraindications to implant surgery (except for type two diabetes in test group).
* Patients irradiated in the head and neck area.
* Immunosuppressed or immunocompromised patients (except for type two diabetes in test group).
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients with untreated periodontitis.
* Patients with poor oral hygiene and motivation.
* Previous guided bone reconstruction at the intended implant sites.
* Uncontrolled diabetes (except for type two diabetes in test group).
* Pregnancy or nursing.
* Substance abuser.
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for implant placement.
* Patients with infection and or inflammation in the area intended for implant placement.
* Patients participating in other studies, if the present protocol cannot be properly adhered to.
* Patients referred only for implant placement and cannot be followed ant the treating centre.
* Patients unable to be followed for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Implant failure | Up to 5 years
  Defined as implant mobility and/or any infection dictating implant removal, and/or implant fracture and/or any other mechanical complication rendering the implant unusable. The stability of each individual implant will be measured by the local blinded outcome assessors manually tightening the screws with a torque of 30 Ncm at abutment connection at initial loading. At 1,3 and 5 years after loading, individual implants will be manually tested for stability. Once the single crowns will be screwed, their stability will be assessed by rocking the crown with the handles of two dental instruments.
Prosthesis failure | Up to 5 years
  Whether it will not be possible to place the prosthesis because of implant failure or a prosthesis that has to be remade for any reason.
Complications | Up to 5 years
  Technical (fracture of the framework and/or the veneering material, screw loosening, etc.) and/or biologic (pain, swelling, suppuration, peri-implantitis, etc.) complications will be considered.

SECONDARY OUTCOMES:
Peri-implant marginal bone level changes | At 1,3 and 5 years
  Peri-implant marginal bone level changes will be assessed on periapical radiographs took with the paralleling technique at implant placement, at initial loading, 1,3 and 5 years after loading. Ideally digital radiographs should be taken, otherwise radiographs on conventional films will be scanned into TIFF format with a 600 dpi resolution, and stored in a personal computer. Peri-implant marginal bone levels will be measured using the Scion Image (Scion Corporation, Frederick, MD, USA) software. The software will be calibrated for every single image using the known distance of the first two consecutive threads. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact. Bone levels will be measured.
Patient satisfaction | At 1,3 and 5 years
  Patients will answer the following questions (separately for each implant):
  Are you satisfied with the function of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  Are you satisfied with the aesthetic outcome of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  Would you undergo the same therapy again? Possible answers: "yes" or "no"
Implant stability quotient (ISQ) | 1,3 and 5 years
  ISQ was measured and recorded using the IS3 (Osstem), at implant placement, at implants exposure, at the impression time, and prosthetic loading.

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Tallarico, Rome, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No